CLINICAL TRIAL: NCT05087927
Title: IGHID 12113 - Formative Study for I'm Fully Empowered4PrEP Intervention on HIV PrEP Uptake by Southern African American Women (IFE4PrEP Formative Study)
Brief Title: Study for IFE4PrEP Intervention on PrEP Uptake by Southern African American Women
Acronym: IFE4PrEP
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-1244
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: HIV Prevention
Keywords: HIV; pre-exposure prophylaxis; PrEP; Prevention; Women's Health; Health Messaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus Group: There will be 4 focus groups of up to 12 women in each focus group.
  Interventions: Behavioral: Gain framing plus demographically targeted photos; Behavioral: Loss framing plus demographically targeted photos; Behavioral: Gain framing plus not demographically targeted photos; Behavioral: Loss framing plus not demographically targeted photos
- Survey Group: There will be up to 200 women who complete the survey for this study.
  Interventions: Behavioral: Gain framing plus demographically targeted photos; Behavioral: Loss framing plus demographically targeted photos; Behavioral: Gain framing plus not demographically targeted photos; Behavioral: Loss framing plus not demographically targeted photos

INTERVENTIONS:
Behavioral: Gain framing plus demographically targeted photos — Gain framing: Participant feels PrEP puts her in control
  Participants (majority of whom will be African American) will be shown an image of women of multiple races.
Behavioral: Loss framing plus demographically targeted photos — Loss framing: Without PrEP, participant feels less in control
  Participants (majority of whom will be African American) will be shown an image of women of multiple races.
Behavioral: Gain framing plus not demographically targeted photos — Gain framing: Participant feels PrEP puts her in control
  Participants (majority of whom will be African American) will be shown an image of an African American woman.
Behavioral: Loss framing plus not demographically targeted photos — Loss framing: Without PrEP, participant feels less in control
  Participants (majority of whom will be African American) will be shown an image of an African American woman.

SUMMARY:
Purpose: This study is partnering with communities to identify the best ways to provide HIV prevention communication and services for women living in public housing who have been disproportionately affected by HIV but underserved by current HIV prevention programs. The investigators want to work with community members to develop and design the delivery of a program to promote awareness of and access to pre-exposure prophylaxis (PrEP) for HIV prevention among women living in public housing.

Participants: Up to 248 cisgender females who are 18 years of age or older and currently reside in Durham Housing Authority (DHA) housing will be enrolled in this study at UNC.

Procedures (methods): Data collection for this formative study will consist of 4 focus groups of up to 12 women in each focus group living in DHA as well as a survey of 200 women living in DHA.

DETAILED DESCRIPTION:
Study Design

This observational formative study consists of cross-sectional data collection with women living in DHA (Durham Housing Authority) housing through surveys and focus group discussions. Both modes of data collection will service to collect descriptive information to refine the intervention. The survey will also include a randomized messaging experiment (see Data Collection Procedures description below).

Study Duration, Enrollment and Number of Subjects

This formative study will last up to one year (12 months). The investigators will enroll up to 248 participants (up to 200 survey participants and up to 48 focus group participants with some women participating in both) as recruitment allows and as necessitated by thematic saturation.

Study Population

The target population for this study is African American cisgender women at least 18 years old residing in DHA community housing. The vast majority of DHA residents are African American, so the investigators anticipate recruiting participants who are majority African American without explicitly excluding prospective participants on the basis of race. Women will be eligible to participate if they meet the following criteria:

1. 18 years of age or older
2. Identify as cisgender female (assigned female sex at birth and currently identify as female)
3. Currently reside in Durham Housing Authority (DHA) housing

Data Collection Procedures

Survey

The self-administered electronic survey will assess the topics listed below and will include a randomized messaging experiment to assess the effect of exposure messaging about PrEP with variable framing on attitudes and perceived norms about PrEP. Participants will complete the survey as follows:

* Women recruited through community network referral may complete the survey on their own device at the time of their choosing.
* Women recruited through community/public events or FGDs will be provided the option to either: a) complete the self-administered electronic survey during the event on a study-owned device (if an in-person event). Limited literacy, vision-impaired, or any participant who desires assistance may request that a study staff member read the questions aloud to them for them to complete the survey, or request to complete the survey as an interviewer-administered survey in a private location; or b) complete the survey at a time of their choosing on their own device.

Survey topics will include:

* Sociodemographic characteristics (age, race/ethnicity, DHA community of residence)
* PrEP awareness & knowledge
* Attitudes toward PrEP
* Randomized messaging experiment (see below)
* Perceived PrEP norms
* Perceived ability to access PrEP
* Barriers and facilitators to using PrEP
* Perceived HIV risk
* HIV risk factors/behaviors
* Likelihood to use PrEP/interest/willingness to use PrEP
* Perceived stigmas

The survey will include an embedded randomized 2 x 2 between-subjects experiment (gain vs. loss framing by intrinsic vs. extrinsic motivation messaging) evaluating the effects of the alternative messaging approaches on intermediate endpoints in Table 3 of the protocol to identify the approaches most associated with positive PrEP attitudes and norms. The experiment will be embedded in a questionnaire administered before focus group sessions to 40 focus group participants and to 160 additional women in study communities (total of 200, 50 per community). During each of the 4 focus groups, the investigators also will explore women's reactions to alternative modes (e.g., flyers, posters, apps, social media) of PrEP messaging.

Hypotheses for each messaging attribute are as follows:

H1: Gain framing will be associated with more positive attitudes and more positive perceived norms about PrEP than loss framing.

* Gain framing: PrEP puts me in control
* Loss framing: Without PrEP, I'm less in control

H2: Demographic targeting will be associated with more positive attitudes and more positive perceived norms about PrEP than non-demographically targeted messaging.

* Demographically targeted: [Image of African American woman]
* Extrinsic framing: [Image of women of multiple races]

Focus Group Discussions (FGDs)

Focus Group participants will be given the option to participate in a focus group by Zoom or in person. Per North Carolina Executive Orders current at the time of data collection, the investigators anticipate that in-person FGDs will be conducted in a private indoor location with sufficient ventilation, 6-foot distancing between participants, and with face masks for both FGD facilitators and participants. Focus groups with limited participants showing up may be converted to individual in-depth interviews. With participant consent, FGDs will be audio-recorded for analysis. Zoom focus groups will be video/audio-recorded with the video deleted and the audio retained directly following the FGD. Focus groups will be led by trained study staff members who will facilitate a discussion on the topics below:

* Current awareness & knowledge of PrEP (including current sources of information about PrEP)
* Attitudes toward PrEP (including any stigmas about PrEP, perceived risk)
* Perceptions of and recommendations for messaging about PrEP use among cisgender women (open-ended then specific reactions)
* Perceptions of and recommendations for messaging about PrEP mobile unit (open-ended then specific reactions)
* Preferences for mobile PrEP unit delivery features (e.g., timing, location, appointment type, delivery of complementary services).
* Best media/modes for providing messages about PrEP and the mobile unit to women in DHA.
* Perceptions of peer networkers, best approach for contacting residents and providing information.
* Barriers and facilitators to using PrEP

ELIGIBILITY:
Inclusion Criteria:

Women will be eligible to participate if they meet the following criteria:

* 18 years of age or older
* Identify as cisgender female (assigned female sex at birth and currently identify as female)
* Currently reside in Durham Housing Authority (DHA) housing

Exclusion Criteria:

Women will not be eligible to participate if they meet the following criteria:

* Younger than 18 years of age
* Do not Identify as cisgender female (assigned female sex at birth and currently identify as female)
* Do not currently reside in Durham Housing Authority (DHA) housing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as cisgender female
Study Population: The target population for this study is African American cisgender women at least 18 years old residing in DHA (Durham Housing Authority) community housing. The vast majority of DHA residents are African American, so the investigators anticipate recruiting participants who are majority African American without explicitly excluding prospective participants on the basis of race.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Modified Jaspal, Lopes, and Maatouk Attitudes toward PrEP Scale (APS) | Baseline
  A subset of the Attitudes toward PrEP Scale (APS) will be used to assess the association between message exposure and attitudes toward pre-exposure prophylaxis (PrEP). This sub-set scale will include nine items rated on a 5-point Likert scale (responses ranging from 1=Strongly Disagree to 5=Strongly Agree). The nine items are a sub-set of the original APS scale and will include four items comprising sub-scale 2, three items comprising sub-scale 3, and two items from sub-scale 1. A mean score will be calculated for each complete sub-scale (2 and 3) ranging from 1-5. Each of the two items from sub-scale 1 will be scored individually, ranging from 1-5. Higher scores indicate more positive attitudes toward PrEP.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Golin, MD, Principal Investigator — UNC-Chapel Hill; Lauren Hill, PhD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No